CLINICAL TRIAL: NCT03537547
Title: Combinatorial Pharmacogenomics Testing in Treatment-Naïve Major Depressive Disorder
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Per sponsor and PI institution discussions
Sponsor: Washington University School of Medicine (Other)
Collaborators: AssureRx Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201609109
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Major Depressive Disorder; Depression; Depressive Disorder; Depressive Episode; Depression, Unipolar
Keywords: treatment naive; major depression; pharmacotherapy; pharmacogenomic; genomics
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to have their study clinician have access to their pharmacogenetic report (provide through the GeneSight Psychotropic tool) in order to make treatment decisions, or to not have access to their report for the first 12 weeks. At Visit 5, Week 12, all participants will receive a copy of their pharmacogenetics report and all clinicians will be unblinded for 'open label' to be able to use the results to guide treatment options for an additional 12 weeks.
Who Masked: Participant, Outcomes Assessor
Masking Description: Coordinators at site are blinded, Sponsor and associates are unblinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GeneSight Psychotropic test (Experimental): Participants randomized to have their study clinician have access to their pharmacogenetic report (provided through the GeneSight Psychotropic tool) in order to make treatment decisions for the first 12 weeks. At Visit 5, Week 12, participants will receive a copy of their pharmacogenetics report and clinicians will continue to be able to use the results to guide treatment options for an additional 12 weeks.
  Interventions: Other: GeneSight Psychotropic test; Drug: FDA-approved antidepressant or antipsychotic treatment
- Treatment As Usual (Active Comparator): Participants randomized to treatment as usual will receive treatment from study clinicians who do not have access to the participant's report for the first 12 weeks. At Visit 5, Week 12, participants will receive a copy of their pharmacogenetics report and clinicians will be unblinded to be able to use the results to guide treatment options for an additional 12 weeks.
  Interventions: Drug: FDA-approved antidepressant or antipsychotic treatment

INTERVENTIONS:
Other: GeneSight Psychotropic test — GeneSight Psychotropic test, developed by AssureRx Health, is a genetic test that analyses pre-selected pharmacokinetics and pharmacodynamics genes and results in a composite phenotype and interpretive report, addressing both safety and efficacy of psychiatric medications.
  Other Names: GeneSight test
  Arms: GeneSight Psychotropic test
Drug: FDA-approved antidepressant or antipsychotic treatment — Participant is treated with medications included in the GeneSight Psychotropic product.

SUMMARY:
This study aims to determine whether the GeneSight Psychotropic test can result in better treatment outcomes for patients with treatment-naive major depressive disorder

DETAILED DESCRIPTION:
Major Depressive Disorder is a chronic psychiatric illness that leads to devastating consequences at the individual and societal levels. Today, the choice of treatment continues to be largely based on subjective factors, primarily the clinician and/or patient's preferences, as well as the individual's history of response to treatment, often tainted by recall bias. Psychiatric medication decisions are even more arbitrary when the subject in question has not had past treatment trials. This often leads to a trial and error process and an increasingly resistant disease with each failed trial. Early implementation of an objective tool designed for tailoring medication choice to an individual may prove highly beneficial in decreasing illness chronicity, individual suffering, and economic burden.

GeneSight Psychotropic test is a pharmacogenomic decision support tool, developed to help clinicians make informed, evidence-based decisions about proper drug selection. Therefore, we propose conducting a randomized, double blind, controlled trial to evaluate the impact of the GeneSight Psychotropic test to guide treatment decisions in patients with treatment-naïve (never having taken medication for depression) Major Depressive Disorder.

This study will involve 6 visits over about 24 weeks where participants will be randomized to have their study clinician have access to their pharmacogenetic report in order to make treatment decisions, or to not have access to their report for the first 12 weeks. At Visit 5, Week 12, all participants will receive a copy of their pharmacogenetics report and all clinicians will be unblinded to be able to use the results to guide treatment options for an additional 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18-65 years of age
2. Treatment-naïve major depressive disorder meeting Diagnostic and Statistical Manual 4th Edition (DSM-IV) criteria, without psychosis
3. Total baseline score on the Quick Inventory Of Depressive Symptomatology Clinician-rated (QIDS-C16) and the Quick Inventory Of Depressive Symptomatology Self-Report (QIDS-SR16) rating scale ≥11
4. Good command of the English language

Exclusion Criteria:

1. Patients with a current diagnosis of schizophrenia
2. Patients with a current diagnosis of schizoaffective disorder
3. Patients with a current diagnosis of bipolar disorder (any type)
4. Currently meeting DSM-IV criteria for significant substance use disorder (exception: nicotine use disorder)
5. A diagnosis of personality disorder that may interfere with the patient's ability to improve on pharmacologic treatment, as determined by study investigator
6. Patients currently receiving electroconvulsive therapy(ECT), deep brain stimulation (DBS) or transcranial magnetic stimulation (TMS) treatment
7. History of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic or euthyroid for 6 months
8. Significant unstable medical condition; life threatening disease; hepatic insufficiency; liver transplant recipient; cirrhosis of the liver; need for therapies that may obscure the results of treatment and/or of the study; malignancy (except basal cell carcinoma) and/or chemotherapy within 1 year prior to screening; malignancy more than 1 year prior to screening must have been local and without metastasis and/or recurrence, and if treated with chemotherapy, without nervous system complications
9. History of gastric bypass surgery
10. Acute suicidal intention and/or in need of immediate hospitalization as judged by the investigator
11. Active psychotic symptoms
12. Currently in an inpatient facility
13. History of prior pharmacogenomic testing
14. Currently pregnant or lactating
15. Inability to provide informed consent
16. Any other factor that in the investigators' judgment may affect patient safety or compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2019-08-19 (Actual)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression change score- Week 8 | Baseline to Week 8
  17-item Hamilton Rating Scale for Depression (HAM-D17) to assess mean change in depressive symptoms severity. Total range of the Hamilton Rating Scale for Depression is 0 to 52, with a greater score being an indication of more severe depressive symptoms.

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression change score- Week 4 | Baseline to end of week 4
  17-item Hamilton Rating Scale for Depression (HAM-D17) to assess mean change in depressive symptoms severity. Total range of the Hamilton Rating Scale for Depression is 0 to 52, with a greater score being an indication of more severe depressive symptoms.
Hamilton Rating Scale for Depression change score- Week 12 | Baseline to end of week 12
  17-item Hamilton Rating Scale for Depression (HAM-D17) to assess mean change in depressive symptoms severity. 17-item Hamilton Rating Scale for Depression (HAM-D17) to assess mean change in depressive symptoms severity. Total range of the Hamilton Rating Scale for Depression is 0 to 52, with a greater score being an indication of more severe depressive symptoms.
Hamilton Rating Scale for Depression change score- Week 24 | Baseline to end of week 24
  17-item Hamilton Rating Scale for Depression (HAM-D17) to assess mean change in depressive symptoms severity. 17-item Hamilton Rating Scale for Depression (HAM-D17) to assess mean change in depressive symptoms severity. Total range of the Hamilton Rating Scale for Depression is 0 to 52, with a greater score being an indication of more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Conway, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States